CLINICAL TRIAL: NCT01225536
Title: A Phase 1 Dose Escalation Study of ARQ 736 in Adult Subjects With Advanced Solid Tumors Harboring BRAF and/or NRAS Mutations
Brief Title: Dose Escalation Study of ARQ 736 in Adult Subjects With Advanced Solid Tumors Harboring BRAF and/or NRAS Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 736-101
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Solid Tumor
Keywords: BRAF mutations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 736 (Experimental)
  Interventions: Drug: ARQ 736

INTERVENTIONS:
Drug: ARQ 736 — Subjects in this study will receive ARQ 736 orally at dose levels specified for their respective dose cohorts. Dosing will begin at 900 mg/day (first cohort) and escalate until the recommended Phase 2 dose or maximum tolerated dose is determined. Cycles will be repeated in four-week (28-day) intervals until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, dose adjustment will be permitted.

SUMMARY:
This is an open-label, Phase 1, dose escalation study of oral ARQ 736 administered to subjects with advanced solid tumors harboring the mutation. The study is designed to explore the safety, tolerability, pharmacokinetics and pharmacodynamics of ARQ 736 and to define a recommended Phase 2 dose of ARQ 736.

DETAILED DESCRIPTION:
Treatment will be initiated at a dose level of 450 mg twice daily (900 mg/daily). All cycles/cohorts of therapy will consist of the oral administration of ARQ 736 twice or four times a day, one hour prior to or two hours after the meal for 28 days continuously. Tumor assessments (CT scan or MRI) will be performed at Baseline, and every two cycles (every eight weeks) thereafter or as otherwise clinically indicated. For early assessment of evidence of biological activity of the tumor PET scan may be performed at Baseline and four weeks from the administration of the first dose of ARQ 736 (approximately Cycle 2 Day1).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent granted prior to initiation of any study-specific procedures
* Male or female subjects of ≥ 18 years of age
* All subjects must be positive for a BRAF and/or NRAS mutation
* Histologically or cytologically confirmed locally advanced, inoperable or metastatic solid tumors
* Failure to respond to at least one prior systemic therapy (including previous treatment with BRAF inhibitors) or to whom standard or curative therapy does not exist
* Life expectancy of greater than three months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors
* Hemoglobin (Hgb) ≥10 g/dl
* Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
* Platelet count ≥100 x 10^9/L
* Total bilirubin ≤1.5 × upper limit of normal (ULN)
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 × ULN (≤5 x ULN for subjects with liver metastases)
* Serum creatinine ≤1.5 × ULN or creatinine clearance >60 mL/min/1.73 m^2 for subjects with creatinine levels above institutional normal
* Left Ventricular Ejection Fraction (LVEF) ≥ the institutional lower limit normal (ILLN)
* Male or female subjects of child-producing potential must agree to use double-barrier contraceptive measures, oral contraception or avoidance of intercourse during the study and for 30 days after the last dose of ARQ 736
* Females of childbearing potential must have a negative serum pregnancy test within seven days prior to the first dose of ARQ 736
* Must agree to have tumor and/or skin (nevi) biopsy at baseline and on Day 15 or Day 22 of Cycle 1. Tumor biopsy will be done if the subject has a lesion for which in the Investigator's opinion a non- or minimally invasive tumor biopsy may be performed. If tumor biopsy is not available, skin (nevi) biopsy should be performed.

Exclusion Criteria:

* Anti-cancer chemotherapy, immunotherapy, or investigational agents within four weeks of the first dose of ARQ 736
* Major surgery or radiotherapy within two weeks of the first dose of ARQ 736
* Brain metastases that are progressing or have been documented to be stable for less than six weeks, or for which systemic corticosteroids are required
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as ARQ 736
* Unable or unwilling to swallow the complete daily dose of ARQ 736
* Significant gastrointestinal disorder(s), in the opinion of the Investigator, (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection)
* History of myocardial infarction (MI) within 6 months of the administration of the first dose of ARQ 736 (MI occurring > 6 months of the first dose of ARQ 736 will be permitted)
* History of congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification within 6 months of the administration of the first dose of ARQ 736
* Previous malignancy within 2 years of the first dose of ARQ 736, except carcinoma in-situ of the cervix
* Concurrent uncontrolled illness, including but not limited to:
* Ongoing or active infection, including human immunodeficiency virus (HIV) infection or bleeding
* Psychiatric illness/substance abuse/social situation that would limit compliance with study requirements
* Blood transfusion within five days prior to blood draw being used to confirm eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of study drug in subjects with advanced solid tumors who have BRAF and/or NRAS mutations | Up to treatment discontinuation + 30 days with an estimated treatment duration of 24 weeks

SECONDARY OUTCOMES:
Assess pharmacokinetic profile | During first cycle of treatment (28 days)
Assess pharmacodynamic activity | During first cycle of treatment (28 days) plus Day 1 of each consecutive cycle with an estimated treatment duration of 24 weeks
Determine preliminary evidence of activity | Up to treatment discontinuation with an estimated treatment duration of 24 weeks
Determine recommended Phase 2 dose | Up to treatment discontinuation with an estimated treatment duration of 24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Los Angeles, California
  - New Haven, Connecticut
  - New Brunswick, New Jersey
- Rozzano, Italy